CLINICAL TRIAL: NCT01466062
Title: Multi-center, Open-label, Uncontrolled Clinical Study of Palivizumab in Japanese Newborns, Infants and Young Children at the Age of 24 Months or Less With Immunocompromised Medical Conditions
Brief Title: Clinical Study of Palivizumab in Japanese Newborns, Infants and Young Children at the Age of 24 Months or Less With Immunocompromised Medical Conditions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: M12-420
Record Dates: First submitted 2011-09-12; First posted 2011-11-07 (Estimated); Results first posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Respiratory Syncytial Virus Infection
Keywords: Immunocompromised medical conditions; Respiratory Syncytial Virus Infection; Infant; Newborn; Young children
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Palivizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Palivizumab (Experimental): 15 mg/kg at 30-day intervals; at least 4 intramuscular injections up to a maximum of 7 intramuscular injections as appropriate for prophylaxis of severe respiratory syncytial virus (RSV) during the RSV season.
  Interventions: Drug: Palivizumab

INTERVENTIONS:
Drug: Palivizumab
  Other Names: ABT-315; Synagis

SUMMARY:
To evaluate safety, efficacy and pharmacokinetics of palivizumab in children at the age of 24 months or less with immunocompromised medical conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of parent or legal guardian who is capable and willing to give written informed consent for his/her newborn, infant or young child to participate this study.
2. Japanese newborn, infant or young child at age of 24 months or less.
3. The subject must meet at least one of the following immunocompromised medical conditions (from [a] to [h]), and must be considered by the investigator to be a suitable candidate to receive prophylactic treatment of palivizumab:

   1. Subject has been diagnosed with combined immunodeficiency (severe combined immunodeficiency, X-linked hyper-immunoglobulin M (IgM) syndrome, etc.), antibody deficiency (X-linked agammaglobulinemia, common variable immunodeficiency, non-X-linked hyper-IgM syndrome, etc.) or other immunodeficiency (Wiskott-Aldrich syndrome, DiGeorge syndrome, etc.) at the time of informed consent, or
   2. Subject has been diagnosed with human immunodeficiency virus infection, or
   3. Subject has been diagnosed with Down syndrome without a current hemodynamically significant congenital heart disease at the time of informed consent (subject must have an experience with persistent respiratory symptom or regular outpatient treatment due to respiratory tract infection prior to current RSV season), or
   4. Subject has a history of post organ transplantation at the time of informed consent, or
   5. Subject has a history of post bone marrow transplantation at the time of informed consent, or
   6. Subject is receiving immunosuppressive chemotherapy at the start of study drug administration, or
   7. Subject is receiving systemic high dose corticosteroid therapy (prednisone equivalents 0.5 mg/kg or more every other day, other than inhaler or topical use) at the start of study drug administration, or
   8. Subject is receiving other immunosuppressive therapy (azathioprine, methotrexate, mizoribine, mycophenolate mofetil, cyclophosphamide, cyclosporine, tacrolimus, cytokine inhibitors, etc.) at the start of study drug administration.

Exclusion Criteria:

1. Subject who meets one of the palivizumab indications already approved in Japan.

   * Subject born at 28 weeks of gestation or less and who is age of 12 months or less at the start of study drug administration.
   * Subject born at 29 - 35 weeks of gestation and who is age of 6 months or less at the start of study drug administration.
   * Subject is age of 24 months or less with a history of bronchopulmonary dysplasia requiring medical management within the 6 months prior to the study drug administration.
   * Subject is age of 24 months or less with a current hemodynamically significant congenital heart disease at the start of study drug administration.
2. Subject requires oxygen supplementation, mechanical ventilation, extracorporeal membrane oxygenation, continuous positive airway pressure or other mechanical respiratory or cardiac support at Screening and at the start of study drug administration.
3. Subject has a current active infection including respiratory syncytial virus infection at Screening and at the start of study drug administration.
4. Subject has a serious concurrent medical condition (hepatic dysfunction, persistent seizure disorder, etc.) except those resulting in an immune deficiency condition or renal failure.
5. Subject has received palivizumab prior to the study drug administration.
6. Subject has received any other investigational agents in the past 3 months or 5 half lives prior to the investigational drug administration (whichever is longer).
7. Subject has a history of an allergic reaction or hypersensitivity to constituents of the study drug.
8. Subject has a history of serious adverse reactions or serious allergic reaction to immunoglobulin products or has a history of hypersensitivity to immunoglobulin products, blood products, or other foreign proteins.
9. Subject whose remaining days of life are expected to be less than one year at the time of informed consent.
10. It will be impossible to collect blood as scheduled from the subject.
11. Subject is considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shigeki Hashimoto, PhD, Study Director — AbbVie
Locations (6):
- Japan (6):
  - Site Reference ID/Investigator# 56847, Hyōgo
  - Site Reference ID/Investigator# 56845, Shimotsuke
  - Site Reference ID/Investigator# 56842, Tokyo
  - Site Reference ID/Investigator# 56844, Tokyo
  - Site Reference ID/Investigator# 56846, Tokyo
  - Site Reference ID/Investigator# 56843, Yokohama

REFERENCES:
- See also: Related info — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Palivizumab: 15 mg/kg at 30-day intervals; at least 4 intramuscular injections up to a maximum of 7 intramuscular injections as appropriate for prophylaxis of respiratory syncytial virus (RSV) during the RSV season.
Period: Overall Study
Arm/Group | Palivizumab
Started | 28
Completed | 26
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Palivizumab
Number analyzed (Participants) | 28
Age Continuous [Mean (Standard Deviation); unit: months] | 14.2 (6.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 17
Region of Enrollment [Number; unit: participants]
  Japan | 28

OUTCOME MEASURES:

1. Primary Outcome: Serum Palivizumab Trough Concentrations at Day 1, Day 31, and Day 121
Description: Serum trough concentrations of palivizumab were assessed at Screening, at Day 31 (30 days after the 1st dose) and Day 121 (30 days after the 4th dose).
Time Frame: Day 1 (Screening), Day 31, Day 121
Population: All participants; n=number of non-missing observations.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Palivizumab
Number analyzed (Participants) | 28
µg/mL
  Day 1 (Screening); n=28 | 0 (0)
  Day 31; n=28 | 59.0 (12.9)
  Day 121; n=26 | 91.8 (40.6)

2. Secondary Outcome: Percentage of Participants Requiring Hospitalization For Respiratory Syncytial Virus (RSV) Infection
Time Frame: From the first administration of palivizumab to 30 days after the last administration of palivizumab. Mean (SD) duration of treatment was 183 (37.29) days.
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Palivizumab
Number analyzed (Participants) | 28
percentage of participants | 0 [0.0 to 12.3]

3. Secondary Outcome: Percentage of Participants Who Required Treatment for Respiratory Syncytial Virus (RSV) Infection
Description: Percentage of participants who required any of the investigated treatments (admission in the intensive care unit [ICU], oxygen supplementation, mechanical ventilation, extracorporeal membrane oxygenation, continuous positive airway pressure and other mechanical respiratory support) for disease caused by RSV infection after the initial dose to 30 days after the last dose of the study drug.
Time Frame: as for outcome 2
Population: All participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Palivizumab
Number analyzed (Participants) | 28
percentage of participants
  Intensive-care unit | 0 [0.0 to 12.3]
  Oxygen supplementation | 0 [0.0 to 12.3]
  Mechanical ventilation | 0 [0.0 to 12.3]
  Extracorporeal membrane oxygenation | 0 [0.0 to 12.3]
  Continuous positive airway pressure | 0 [0.0 to 12.3]
  Other mechanical respiratory support | 0 [0.0 to 12.3]

4. Secondary Outcome: Duration of Hospitalization Caused by Respiratory Syncytial Virus (RSV) Infection
Description: Number of days of hospitalization caused by RSV infection.
Time Frame: as for outcome 2
Population: Number of participants hospitalized. Since no subject had a RSV infection from the first administration of palivizumab to 30 days after the administration of palivizumab, the number of participants analyzed was 0 for this measure.
Arm/Group | Palivizumab
Number analyzed (Participants) | 0

5. Secondary Outcome: Duration of Required Treatment for Respiratory Syncytial Virus (RSV) Infection
Description: Duration (days) of requirement for any of the investigated treatments (admission in the intensive care unit [ICU], oxygen supplementation, mechanical ventilation, extracorporeal membrane oxygenation, continuous positive airway pressure and other mechanical respiratory support) for disease caused by RSV infection after the initial dose to 30 days after the last dose of the study drug.
Time Frame: as for outcome 2
Population: Number of participants who required any of the investigated treatments for RSV. Since no subject had a RSV infection from the first administration of palivizumab to 30 days after the administration of palivizumab, the number of participants analyzed was 0 for this measure.
Arm/Group | Palivizumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and Discontinuations Due to AEs
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with treatment. If an adverse event meets any of the following criteria, it is considered a serious adverse event (SAE): results in death or is life-threatening, results in admission or prolongation of hospitalization, results in congenital anomaly or persistent or significant disability/incapacity, or is an important medical event requiring medical or surgical intervention to prevent serious outcome. AEs were categorized by severity (mild, moderate, severe) and relationship to treatment (probably, possibly, probably not, not related). Please see Adverse Events section below for more details.
Time Frame: From the first administration of palivizumab to 100 days after the last administration of palivizumab. Mean (SD) duration of treatment was 183 (37.29) days.
Population: All participants
Measure: Number; unit: participants
Arm/Group | Palivizumab
Number analyzed (Participants) | 28
participants
  Any AE | 27
  Any AE at least "possibly" drug related | 0
  Any AE at least "probably not" drug related | 7
  Any "severe" AE | 2
  Any SAE | 7
  Any AE leading to discontinuation of study drug | 1
  Any AE leading to death | 0
  Death | 0

7. Secondary Outcome: Mean Baseline and Mean Change From Baseline in Systolic/Diastolic Blood Pressure at Day 121
Time Frame: Baseline (Day 1), Day 121 (30 days after the 4th dose)
Population: All participants; n= number of participants with measurements at given time points.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Palivizumab
Number analyzed (Participants) | 28
mm Hg
  Baseline Systolic Blood Pressure (SBP); n=26 | 96.1 (9.44)
  Change from Baseline in SBP at Day 121; n=26 | -2.4 (10.23)
  Baseline Diastolic Blood Pressure (DBP); n=25 | 55.0 (9.16)
  Change from Baseline in DBP at Day 121; n=25 | 3.0 (14.56)

8. Secondary Outcome: Mean Baseline and Mean Change From Baseline in Body Temperature at Day 121
Time Frame: Baseline (Day 1), Day 121 (30 days after the 4th dose)
Population: All participants with measurements at given time points.
Measure: Mean (Standard Deviation); unit: degrees Celcius
Arm/Group | Palivizumab
Number analyzed (Participants) | 26
degrees Celcius
  Baseline Body Temperature (BT) | 36.77 (0.346)
  Change from Baseline in BT at Day 12 | -0.11 (0.400)

9. Secondary Outcome: Mean Baseline and Mean Change From Baseline in Respiratory Rate at Day 121
Time Frame: Baseline (Day 1), Day 121 (30 days after the 4th dose)
Population: All participants with measurements at given time points.
Measure: Mean (Standard Deviation); unit: respirations per minute
Arm/Group | Palivizumab
Number analyzed (Participants) | 26
respirations per minute
  Baseline Respiratory Rate (RR) | 33.4 (8.59)
  Change from Baseline in RR at Day 121 | 1.5 (8.21)

10. Secondary Outcome: Mean Baseline and Mean Change From Baseline in Pulse Rate at Day 121
Time Frame: Baseline (Day 1), Day 121 (30 days after the 4th dose)
Population: All participants with measurements at given time points.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Palivizumab
Number analyzed (Participants) | 26
beats per minute
  Baseline Pulse Rate (PR) | 126.6 (21.91)
  Change from Baseline PR at Day 121 | -6.7 (26.66)

11. Secondary Outcome: Mean Baseline and Mean Change From Baseline in Body Weight at Day 121
Time Frame: Baseline (Day 1), Day 121 (30 days after the 4th dose)
Population: All participants with measurements at given time points.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Palivizumab
Number analyzed (Participants) | 26
kilograms
  Baseline Body Weight (BW) | 8.76 (1.90)
  Change from Baseline in BW at Day 121 | 1.23 (0.71)

12. Secondary Outcome: Hematology: Mean Baseline and Mean Change From Baseline in Hemoglobin at Day 121
Description: Normal range for hemoglobin varied by the monthly age of the participant.
Time Frame: Baseline (Day 1), Day 121 (30 days after the 4th dose)
Population: All participants with measurements at given time points.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Palivizumab
Number analyzed (Participants) | 25
g/dL
  Baseline Hemoglobin | 11.57 (1.56)
  Change from Baseline in Hemoglobin at Day 121 | 0.14 (1.87)

13. Secondary Outcome: Hematology: Mean Baseline and Mean Change From Baseline in Hematocrit at Day 121
Description: Normal range for hematocrit varied by the monthly age of the participant.
Time Frame: Baseline (Day 1), Day 121 (30 days after the 4th dose)
Population: All participants with measurements at given time points.
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | Palivizumab
Number analyzed (Participants) | 25
percentage of red blood cells
  Baseline Hematocrit | 34.32 (4.72)
  Change from Baseline in Hematocrit at Day 121 | 0.96 (5.43)

14. Secondary Outcome: Hematology: Mean Baseline and Mean Change From Baseline in White Blood Cells (WBC), Neutrophils, Eosinophils, Basophils, Lymphocytes, and Monocytes at Day 121
Description: Normal ranges for WBC, neutrophils, eosinophils, basophils, lymphocytes, and monocytes varied by the monthly age of the participant.
Time Frame: Baseline (Day 1), Day 121 (30 days after the 4th dose)
Population: All participants; n=number of participants with measurements at given time points.
Measure: Mean (Standard Deviation); unit: cells *10^3/µL
Arm/Group | Palivizumab
Number analyzed (Participants) | 28
cells *10^3/µL
  Baseline White Blood Cells (WBC); n=25 | 6.74 (3.93)
  Change from Baseline in WBC at Day 121; n=25 | 0.24 (2.53)
  Baseline (BL) Neutrophils; n=24 | 2.60 (2.17)
  Change from BL in Neutrophils at Day 121; n=24 | -0.05 (1.60)
  Baseline Eosinophils; n=24 | 0.25 (0.26)
  Change from BL in Eosinophils at Day 121; n=24 | -0.0 (0.31)
  Baseline Basophils; n=24 | 0.04 (0.05)
  Change from Baseline in Basophils at Day 121; n=24 | 0.02 (0.07)
  Baseline Lymphocytes; n=24 | 3.36 (2.35)
  Change from BL in Lymphocytes at Day 121; n=24 | 0.31 (1.69)
  Baseline Monocytes; n=24 | 0.51 (0.44)
  Change from Baseline in Monocytes at Day 121; n=24 | -0.02 (0.38)

15. Secondary Outcome: Hematology: Mean Baseline and Mean Change From Baseline in Red Blood Cells (RBC) and Platelet Count at Day 121
Description: Normal ranges for RBC and platelet count varied by the monthly age of the participant.
Time Frame: Baseline (Day 1), Day 121 (30 days after the 4th dose)
Population: All participants with measurements at given time points.
Measure: Mean (Standard Deviation); unit: cells *10^4/µL
Arm/Group | Palivizumab
Number analyzed (Participants) | 25
cells *10^4/µL
  Baseline Red Blood Cells (RBC) | 410.6 (70.83)
  Change from Baseline in RBC at Day 121 | 22.3 (74.74)
  Baseline Platelet Count | 31.29 (19.80)
  Change from Baseline in Platelet Count at Day 121 | 1.72 (18.35)

16. Secondary Outcome: Blood Chemistry: Mean Baseline and Change From Baseline in Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), and Alanine Aminotransferase (ALT) at Day 121
Description: Normal ranges for ALP, AST, and ALT varied by the monthly age of the participant.
Time Frame: Baseline (Day 1), Day 121 (30 days after the 4th dose)
Population: All participants with measurements at given time points.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Palivizumab
Number analyzed (Participants) | 24
U/L
  Baseline ALP | 943.0 (519.10)
  Change from Baseline in ALP at Day 121 | -18.0 (368.35)
  Baseline AST | 39.08 (12.95)
  Change from Baseline in AST at Day 121 | 1.54 (8.09)
  Baseline ALT | 31.13 (25.70)
  Change from Baseline in ALT at Day 121 | -3.17 (14.07)

17. Secondary Outcome: Blood Chemistry: Mean Baseline and Change From Baseline in Total Bilirubin, Blood Urea Nitrogen (BUN), Creatinine, and C-reactive Protein (CRP) at Day 121
Description: Normal ranges for total bilirubin, BUN, creatinine, and CRP varied by the monthly age of the participant.
Time Frame: Baseline (Day 1), Day 121 (30 days after the 4th dose)
Population: All participants with measurements at given time points.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Palivizumab
Number analyzed (Participants) | 24
mg/dL
  Baseline Total Bilirubin | 0.30 (0.14)
  Change from Baseline in Total Bilirubin at Day 121 | 0.04 (0.15)
  Baseline BUN | 11.46 (4.52)
  Change from Baseline in BUN at Day 121 | 0.87 (4.64)
  Baseline Creatinine | 0.23 (0.04)
  Change from Baseline in Creatinine at Day 121 | 0.01 (0.04)
  Baseline CRP | 0.29 (0.42)
  Change from Baseline in CRP at Day 121 | 0.03 (0.62)

18. Secondary Outcome: Urinalysis: Presence of Urine Protein, Glucose, and Occult Blood at Screening and Day 121
Description: The values -, -/+, 1+, 2+, 3+, and 4+ represent a range from none (-) to highest (4+) presence of protein, glucose, and occult blood in the urine. Table presents the number of participants with each value. Those categories with 0 participants to report at either time point are not included in the table below.
Time Frame: Screening, Day 121 (30 days after the 4th dose)
Population: All participants; n=number of participants with measurements at given time points.
Measure: Number; unit: participants
Arm/Group | Palivizumab
Number analyzed (Participants) | 28
participants
  Protein "-" at Screening; n=24 | 21
  Protein "+/-" at Screening; n=24 | 3
  Protein "-" at Day 121; n=22 | 21
  Protein "+/-" at Day 121; n=22 | 1
  Glucose "-" at Screening; n=24 | 24
  Glucose "-" at Day 121; n=22 | 22
  Occult Blood "-" at Screening; n=24 | 21
  Occult Blood "+/-" at Screening; n=24 | 2
  Occult Blood "1+" at Screening; n=24 | 1
  Occult Blood "-" at Day 121; n=22 | 21
  Occult Blood "+/-" at Day 121; n=22 | 0
  Occult Blood "1+" at Day 121; n=22 | 1

ADVERSE EVENTS:
Time Frame: AEs:from time of initial study drug administration (Day 1) to 100 days after final administration of the study drug. SAEs:from screening period until 100 days after final administration of study drug. Mean (SD) duration of treatment was 183 (37.29) days.
Arm/Group | Palivizumab
Serious Adverse Events (participants affected / at risk) | 7/28
Other Adverse Events (participants affected / at risk) | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palivizumab (N=28)
Duodenal Stenosis (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastrointestinal Perforation (Gastrointestinal disorders) | 1
Bronchitis (Infections and infestations) | 2
Croup Infectious (Infections and infestations) | 1
Infectious Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia Bacterial (Infections and infestations) | 1
Encephalopathy (Nervous system disorders) | 1
Gastroenteritis (Infections and infestations) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palivizumab (N=28)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Hypercoagulation (Blood and lymphatic system disorders) | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Antithrombin III Deficiency (Congenital, familial and genetic disorders) | 1
Conjunctivitis (Eye disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Mouth Haemorrhage (Gastrointestinal disorders) | 1
Rectal Prolapse (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 3
Hepatic Function Abnormal (Hepatobiliary disorders) | 4
Hypogammaglobulinaemia (Immune system disorders) | 5
Bronchitis (Infections and infestations) | 4
Conjunctivitis Infective (Infections and infestations) | 1
Cystitis (Infections and infestations) | 2
Exanthema Subitum (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 7
Gastroenteritis Viral (Infections and infestations) | 1
Impetigo (Infections and infestations) | 1
Influenza (Infections and infestations) | 6
Molluscum Contagiosum (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 5
Otitis Media (Infections and infestations) | 2
Otitis Media Acute (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 3
Pseudomonas Infection (Infections and infestations) | 1
Respiratory Tract Infection (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Rotavirus Infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tinea Cruris (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 10
Upper Respiratory Tract Infection Bacterial (Infections and infestations) | 1
Viral Infection (Infections and infestations) | 1
Arthropod Sting (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Radiation Skin Injury (Injury, poisoning and procedural complications) | 1
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 1
Thermal Burn (Injury, poisoning and procedural complications) | 1
Antithrombin III Decreased (Investigations) | 1
Bacterial Test Positive (Investigations) | 1
C-Reactive Protein Increased (Investigations) | 2
Neutrophil Count Decreased (Investigations) | 1
Neutrophil Count Increased (Investigations) | 1
White Blood Cell Count Increased (Investigations) | 1
White Blood Cells Urine Positive (Investigations) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Febrile Convulsion (Nervous system disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 2
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 9
Eczema Asteatotic (Skin and subcutaneous tissue disorders) | 4
Eczema Infantile (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis Palmaris And Plantaris (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 5
Urticaria (Skin and subcutaneous tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 4
Constipation (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.